CLINICAL TRIAL: NCT03494907
Title: A Randomized, Double-blind, Placebo- and Positive-controlled, Single-dose, 4-way Crossover Study to Evaluate the Effects of Seltorexant (JNJ-42847922) on Electrocardiogram Intervals in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effects of Single-dose Seltorexant on Electrocardiogram Intervals in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CR108459; 2017-004770-33 (EudraCT Number); 42847922MDD1007 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-04-05; First posted 2018-04-11 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Seltorexant (Low and high dose) (Experimental): Participants will receive seltorexant tablets orally in 2 of 4 treatment arms (A,B,C,D) in a cross-over design, with 7 days wash-out phase between each treatment period.
  Interventions: Drug: Seltorexant
- Moxifloxacin (Experimental): Participants will receive moxifloxacin tablets orally in 1 of 4 treatment arms (A,B,C,D) in a cross-over design, with 7 days wash-out phase between each treatment period.
  Interventions: Drug: Moxifloxacin Dose 1
- Placebo Matched to Seltorexant (Experimental): Participants will receive seltorexant placebo tablets orally in 3 of 4 treatment arms (A,B,C,D) in a cross-over design, with 7 days wash-out phase between each treatment period.
  Interventions: Other: Placebo Matched to Seltorexant
- Placebo Matched to Moxifloxacin (Experimental): Participants will receive moxifloxacin placebo tablets orally in 3 of 4 treatment arms (A,B,C,D) in a cross-over design, with 7 days wash-out phase between each treatment period.
  Interventions: Other: Placebo Matched to Moxifloxacin

INTERVENTIONS:
Drug: Seltorexant — Participants will be administered oral dose of seltorexant over-encapsulated tablets on Day 1.
  Other Names: JNJ-42847922
  Arms: Seltorexant (Low and high dose)
Other: Placebo Matched to Seltorexant — Participants will be administered matching placebo to seltorexant tablets on Day 1.
  Arms: Placebo Matched to Seltorexant
Other: Placebo Matched to Moxifloxacin — Participants will be administered oral dose of moxifloxacin placebo tablet on Day 1.
  Arms: Placebo Matched to Moxifloxacin
Drug: Moxifloxacin Dose 1 — Participants will be administered oral dose 1 of moxifloxacin on Day 1.
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to assess the effects of single dose seltorexant on QT/QTc intervals and electrocardiogram (ECG) morphology at therapeutic and supratherapeutic exposures in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Have signed informed consent form (ICF) indicating they understand the purpose of and procedures required for the study, including the required pharmacogenomic component (which specifies testing of genes predisposing to long or short QT and related cardiac syndromes), and are willing to participate in the study. Consent for sample storage will be obtained in the ICF
* Be Willing to adhere to the prohibitions and restrictions specified in the protocol
* A female participant must be either not of childbearing potential (ie, postmenopausal, permanently sterile) or of childbearing potential and practicing a highly effective method of contraception (failure rate of less than [<]1 percent [%] per year when used consistently and correctly)
* A female participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study drug administration
* A male participant, who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. Heart rate between 45 and 100 beats per minute (bpm), inclusive

Exclusion Criteria:

* Clinically significant abnormal values for hematology, serum chemistry (including thyroid stimulating hormone [TSH] at screening only) or urinalysis at screening or at admission to the study site
* Clinically significant abnormal physical examination, vital signs, or 12-lead electrocardiogram (ECG) at screening or at admission to the study site as deemed appropriate by the investigator
* Received a known inhibitor of CYP3A4 or CYP2C9 activity within 14 days or a period less than 5 times the drugs' half-life; whichever is longer, before the first dose of the study drug is scheduled
* Known allergy to the study drug or any of the excipients of the formulation
* Received an experimental drug or used an experimental medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before the first dose of the study drug is scheduled
* A woman who is pregnant, breast-feeding, or planning to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in QT/QTc Intervals | Baseline up to Day 3
  Change from baseline in QT and QTc interval will be assessed. QT interval will be measured in triplicates from 12 lead Holter extracted triplicate ECG recordings and corrected QT (QTc) interval will be calculated based on Fridericia (QTcF), Bazett (QTcB), and/or study specific power (QTcP) equations.
Percentage of Participants with Change from Baseline in T-wave Morphology | Baseline up to Day 3
  The percentage of participants in each treatment having T-wave morphology changes from baseline that represent the appearance or worsening of the morphological abnormality will be reported.
Percentage of Participants with Change from Baseline in U-wave Morphology | Baseline up to Day 3
  The percentage of participants with change from baseline with abnormal U-waves morphology that represent the appearance or worsening of the morphological abnormality will be reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  Cmax is the maximum observed plasma concentration of seltorexant and its circulating metabolites.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  Tmax is the time to reach the maximum observed plasma concentration of seltorexant and its circulating metabolites.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration of seltorexant and its circulating metabolites.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant. AUC (0-infinity) will be assessed for seltorexant and its circulating metabolites.
Elimination Half-Life (t1/2) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).
Total Apparent Clearance (CL/F) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  CL/F for extravascular administration divided by the fraction of dose absorbed, calculated using the observed value of the last non-zero plasma concentration.
Apparent Volume of Distribution (Vd/F) | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Metabolite to Parent (M/P) Ratio for AUC[last] | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  M/P Ratio AUC[last] is the ratio of AUC[last] of seltorexant to AUC[last] of seltorexant's metabolites.
Metabolite to Parent (M/P) Ratio for AUC[infinity] | Pre-dose; 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours Post-dose
  M/P Ratio AUC[infinity] is the ratio of AUC[infinity] of seltorexant to AUC[infinity] of seltorexant's metabolites.
Relationship Between the Plasma Concentrations of Seltorexant and Changes in the QT/QTc Interval | Up to Day 3
  The relationship between change in QT/QTc interval and plasma concentrations from both doses of seltorexant at matching time points will be assessed.
Number of Participants with Adverse Events and Serious Edverse Events as a Measure of Safety and Tolerability | Approximately 11 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium